CLINICAL TRIAL: NCT05084118
Title: A Prospective, Randomized, Double- Blind, Placebo- Controlled Study to Evaluate the Efficacy of Landiolol Hydrochloride for Prevention of Atrial Fibrillation in Patients Undergoing Cardiac Surgery
Brief Title: Landiolol for Prevention of Postoperative Atrial Fibrillation in Patients Undergoing Cardiac Surgery
Acronym: LANDI-POAF
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Andreas Binder, Prinicipal Investigator, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LAN_POAF_01
Record Dates: First submitted 2021-05-18; First posted 2021-10-19 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Atrial Fibrillation; Postoperative Complications
Keywords: landiolol
MeSH Terms: conditions — Atrial Fibrillation; Postoperative Complications

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Landiolol group (Active Comparator): Randomized patients receiving low dose landiolol after cardiac surgery
  Interventions: Drug: Landiolol HCl
- Placebo group (Placebo Comparator): Randomized patients receiving 0,9% saline solution after cardiac surgery
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Landiolol HCl — continous 2mcg/kg/min low dose application of Landiolol HCl for 72 hours
  Other Names: Rapibloc
  Arms: Landiolol group
Drug: Placebo — continous application of isotone saline solution for 72 hours
  Other Names: Isotone saline solution
  Arms: Placebo group

SUMMARY:
Postoperative atrial fibrillation (POAF) is the most common arrhythmia after cardiac surgery with incidences ranging from 20% to 40% with the consequence of increasing mortality, morbidity, and hospital length of stay, as well as increasing the costs to the health care system. To prevent POAF the use of beta-blockers is suggested by the EACTA and ESC guidelines. Despite the prophylactic use, the discontinuation of beta-blockers in the perioperative period is a known risk factor that contributes to the occurrence of POAF. Due to the short half time and the highly beta-1-selective properties of Landiolol, it could be possible to initiate a betablocker for prevention in the immediate postoperative setting, without adverse effects like hypotension or severe bradycardia as seen with other betablockers like Metoprolol or even sometimes Esmolol.

Landiolol is already approved for the treatment of atrial tachycardias but is not yet approved for the use of prevention of POAF. In multiple previous studies the preventive potential of Landiolol in cardiac surgery could be proven in japanese study populations, with limitations due to limited sample sizes. In these trials the use of low-dose Landiolol effectively reduced the incidence of POAF without significant differences of increased side effects or in the hemodynamic stability compared to the placebo or standard of care groups.

The primary objective of this prospective, double-blind, randomized, placebo-controlled phase III trial is to prove that the postoperative application of low-dose Landiolol significantly reduces the incidence of POAF without increased adverse events or hemodynamic instability compared to the placebo group after cardiac surgery in a non-Asian population.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥ 18 years old
2. Written informed consent from patient
3. Patients are in sinus rhythm
4. Oral Betablocker in the patients long-term medication
5. One of the following cardiac surgical procedures which is planned on cardiopulmonary bypass (CPB):

   1. Single valve surgery
   2. Single or multiple CABG procedures
   3. Single valve surgery in combination with one or multiple coronary artery bypass grafts (CABGs)
   4. Multiple valve surgery in combination with or without CABG
   5. Single or multiple valve surgery in combination with ascending aorta procedure with or without additional CABG
   6. Re-surgery of aortic valve, mitral valve, aortic arch or ascending aorta with or without CABG
6. Cardiac surgery is performed electively

Exclusion Criteria:

1. Bodyweight > 101kg and/or BMI ≥ 40
2. Cardiac surgery is planned as minimally invasive procedure (e.g., without thoracotomy or with lateral incision, minimal thoracotomy) or planned as off-pump surgery
3. Planned maze procedure, radiofrequency ablation, pulmonary vein ablation, resection of the atrial appendix or atrial resections during the surgery
4. Sinus bradycardia (resting heart rate < 50/min) at screening and before start of IMP treatment
5. Second- or third-degree atrioventricular block at screening and before start of IMP treatment
6. Clinical hypothyroidism or hyperthyroidism at screening
7. History of ventricular arrhythmia
8. Permanent atrial fibrillation or atrial fibrillation at time of screening and IMP administration
9. Emergency cardiac surgery
10. Requiring inotropic, vasopressor or requiring ventilatory support at time of screening
11. Circulatory shock requiring mechanical circulatory support before initiation of study medication
12. Distributive shock (cardiac index>2.2 L/min with norepinephrine dose > 0.3 µg/kg/min to reach mean arterial pressure > 65mmHg) before initiation of study medication
13. More than 5 units of RBC necessary to maintain a haemoglobin level >8mg/dl at the end of surgery
14. Prior cardiac surgery within the past 6 months
15. History of heart transplantation or planned heart transplantation
16. Any other disease or condition that is likely to interfere with the evaluation of the study drug, outcome assessment or satisfactory conduct of the study:

    1. Active infective endocarditis
    2. Stroke or transient ischemic attack (TIA) within the last 6 months
    3. Concomitant disease with a life expectancy of less than 6 months
    4. Cardiopulmonary resuscitation within the last 4 weeks
    5. Patients requiring renal replacement therapy
17. Active infection on current systemic antibiotics and/ or temperature greater than 38°C at time of screening and before start of surgery
18. Haemoglobin < 5 mmol/l (< 8.06 g/dl)
19. Any systemic anti-cancer therapy within past 3 months
20. Patients with known hypersensitivity to any constituent of the IMP
21. General exclusion criteria:

    1. Pregnant (in women of childbearing potential a urine or blood pregnancy test has to be performed) or breast-feeding women. Women with childbearing potential (defined as within two years of their last menstruation) not willing to practice appropriate contraceptive measures (e.g., implanon, injections, oral contraceptives, intrauterine devices, partner with vasectomy, abstinence) while participating in the trial
    2. Participation in any interventional clinical trial within the last one-month prior randomization in this clinicaltrial (screening failures can be rescreened, if appropriate)
    3. Alcohol, drug, or medication abuse
    4. Employee at the study site, spouse/partner or relative of any study staff (e.g., investigator, subinvestigators, or study nurse) or relationship to the sponsor

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2021-10-21 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
The primary end point is a combined endpoint consisting of the occurrence of atrial fibrillation and mortality during the initial 72 hours period after surgery | 3 days
  Death from any reason or the occurence of atrial in the holter ecg within 3 days after operation.

SECONDARY OUTCOMES:
Incidence/ frequency of occurrence of atrial fibrillation during the first seven days after cardiac surgery | 7 days
  The occurence of AF in the holter ecg in the 7 days after the operation
Hemodynamic stability during treatment with IMP | 7 days
  Hemodynamic stability assessed with the need for vasoactive medication in the two groups within 7 days after operation
Length of ICU stay | 30 days
  Postoperative length of stay in days in the icu
Requirement of intensive respiratory and circulatory support | 30 days
  Length of invasive ventilation in hours or need for circulatory support
Peri- and postoperative mortality | 30 days
  Peri- and postoperative mortality
Assessment of biomarkers as surrogate parameters for cardiac dysfunction | 30 days
  Assessment of cardiac biomarkers to evaluate cardiac dysfunction
Biomarker Assessment for cardiac injury, remodelling and fibrosis | 7 days
  Biomarker assessment (TropT, CK, CK-MB, sST-2) for cardiac remodelling, fibrosis, apoptosis and ischemia reperfusion injury at time of start of the surgery, at ICU admission, 24 hours after ICU admission, 3 days and 7 days after surgery.
Incidence of serious adverse events | 30 days
  Incidence of serious adverse events
Echocardiographic assessment for left ventricular function | 7 days
  Echocardiographic assessment for left ventricular systolic, diastolic and valvular function 7 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Binder, Principal Investigator — Medical University of Vienna, Division of Cardiothoracic and Vascular Anesthesia
Locations (1):
- University Hospital Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided